CLINICAL TRIAL: NCT02580084
Title: Prospective Randomized Clinical Study of the Aorta-femoral Bypass and Hybrid Intervention and the Iliac Arteries With Stenting and Plasty of the Common Femoral Artery Effectiveness in Patients With the Iliac Segment and Femoral Artery Occlusive Disease (TASC C, D)
Brief Title: Clinical Study of the Aorta-femoral Bypass and Hybrid Intervention and the Iliac Arteries With Stenting and Plasty of the Common Femoral Artery Effectiveness in Patients With the Iliac Segment and Femoral Artery Occlusive Disease (TASC C, D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NRICP111
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-05

CONDITIONS: Atherosclerosis of the Peripheral Arteries
Keywords: atherosclerosis of the peripheral arteries; Aorta-femoral Bypass; Hybrid Intervention; Iliac Arteries With Stenting and Plasty of the Common Femoral Artery; plastic arteries with lesions of the common femoral artery and deep femoral artery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- aorta femoral bypass (Active Comparator): It is sufficient to identify only the anterior-lateral aorta surface. After heparinization the aorta is clamped above and below the anastomosis. The aorta is dissected along the anterior wall, calcium portions or mural thrombus are removed. Prosthesis is cut obliquely and anastomosis suturing starts with distal angle. Occluded at the prosthetic base jaws, aortic compressor is removed, restoring blood flow in the lower limb. Next stage is tunnel creating for jaws prosthesis conduction on hip. Ureters must remain over the prosthesis, jaw should be above the iliac arteries. After jaws prosthesis conduction on hip distal anastomosis is formed with twisting controlling. Before anastomosis completion the testing jaws and all arteries bloodletting is performed.
  Interventions: Procedure: Aorta femoral Bypass
- hybrid intervention (Experimental): Iliac Arteries With Stenting and Plasty of the Common Femoral Artery
  Interventions: Procedure: Hybrid Intervention

INTERVENTIONS:
Procedure: Hybrid Intervention — The puncture of the femoral artery general is executed and the introducer 7Fr is set. Further, the hydrophilic conductor executes a recanalization of the Vasa of iliac artery occlusion. if you cannot pass the occlusion retrograde is additional access to antegrade recanalization. Then using hydrophilic conductors, an iliac artery antegrade or retrograde recanalization of the Vasa is made.
  Femoral artery arteriotomy. Further execute a direct endarterectomy femoral artery and from the mouth of a hip artery.
  arteriotomy of the femoral artery is closed with a vascular patch use (synthetic or biological).
  Balloon angioplasty and stenting, iliac artery is done, the controlling angiography Closing maims.
  Arms: hybrid intervention
Procedure: Aorta femoral Bypass — It is sufficient to identify only the anterior-lateral aorta surface. After heparinization the aorta is clamped above and below the anastomosis. The aorta is dissected along the anterior wall, calcium portions or mural thrombus are removed. Prosthesis is cut obliquely and anastomosis suturing starts with distal angle. Occluded at the prosthetic base jaws, aortic compressor is removed, restoring blood flow in the lower limb. Next stage is tunnel creating for jaws prosthesis conduction on hip. Ureters must remain over the prosthesis, jaw should be above the iliac arteries. After jaws prosthesis conduction on hip distal anastomosis is formed with twisting controlling. Before anastomosis completion the testing jaws and all arteries bloodletting is performed.
  Arms: aorta femoral bypass

SUMMARY:
Currently, according to the TASC II consensus document (2007) and the Russian guidelines for limb ischemia treatment (2010), aorta-iliac C and D type segment lesions the open surgery is suggested.

DETAILED DESCRIPTION:
Currently, according to the TASC II consensus document (2007) and the Russian guidelines for limb ischemia treatment (2010), aorta-iliac C and D type segment lesions the open surgery is suggested.

According to different studies, 76% occlusive aorta-iliac article course patients indicate femoral-popliteal segment lesions. Due to the lack of inflow and outflow ways of correction needed for adequate limb revascularization surgery treatment of multistorey atherosclerotic lesions patients is still one of the most complex problems of vascular surgery. Perioperational mortality of critical limb ischemia patients reaches 5-10% in retrograde aorta-iliac segment reconstruction.

Due to its high efficiency hybrid operative invasion is one of the most perspective directions in reconstructive vascular surgery development (92-98% of the cases with the small number of post-operative complications).

Furthermore, hybrid surgery is possible with the critical iliac segment and femoral artery lesions, since stenting in the field of physiological bends (femoral artery) may lead to its breaking and artery thrombosis. Arterial segments blood flow reconstruction is possible with hybrid innervations meaning iliac segment stenting and common femoral artery patch.

All reports of iliac arteries stenosis percutaneous angioplasty indicate that the primary technical and clinical success rate exceeds 90%. The technical success of iliac arteries long occlusions recanalization reaches 80-85%. Improvement of endovascular equipment designed for the total occlusions treatment increases technical success of recanalization. The TASC II materials summarize the several large studies results which present the data on the operated segment artery patency at the level of 70-81% within 5-8 years of follow up. A large number of authors note the actuality of aortic-iliac type C and D segment lesions endovascular treatment recommendations revision according to the TASC II, together with hybrid technics implementation in this category of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of C and D type iliac segment and steno-occlusive lesions of the common femoral artery, and with chronic lower limb ischemia (II-IV degree by Fontaine, 2-5 degree by Rutherford), age: 47-75 years old.
* Patients who consented to participate in this study

Exclusion Criteria:

* Chronic heart failure of III-IV functional class by New York Heart Association classification.
* Patients who have suffered a stroke or myocardial infarction less than 3 months
* Significant Steno-occlusive lesion of the contralateral side
* Decompensated chronic "pulmonary" heart
* Aortoarteritis
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy
* Cancer in the terminal stage with a life expectancy less than 6 months
* Expressed aortic calcification tolerant to angioplasty
* Patient refusal to participate or continue to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Safety assessment in the 30-day period: clinically significant bleeding, hematoma, infection of the prosthesis, infection of the postoperative wound, lymphorrhea, renal failure, myocardial infarction, stroke, mortality, thrombosis of the operated segment | 30 days
  Identification of serious adverse events requiring correction of therapy or surgery. Will be used physiological parameter and questionnaire. Classification of bleeding will be used GUSTO (Severe or moderate)
Evaluation of efficiency: primary patency, secondary patency success of procedures, length of hospital stay | 30 days
  If a damage confirmed by duplex is detected, repeat intervention is performed on the side of the examined segment
Evaluation of efficiency: success of procedures | 30 days
  Technical feasibility of the procedure

SECONDARY OUTCOMES:
mortality | during the whole period of observation. Observation is 36 month after surgery
stroke | during the whole period of observation. Observation is 36 month after surgery
myocardial infarction | during the whole period of observation. Observation is 36 month after surgery
limb salvage | in the early postoperative period. Surveillance is 36 month after surgery
infection of the prosthesis | during the whole period of observation. Observation is 36 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NRICP, Novosibirsk, Russia

REFERENCES:
- [Derived] Starodubtsev V, Mitrofanov V, Ignatenko P, Gostev A, Preece R, Rabtsun A, Saaya S, Popova I, Karpenko A. Editor's Choice - Hybrid vs. Open Surgical Reconstruction for Iliofemoral Occlusive Disease: A Prospective Randomised Trial. Eur J Vasc Endovasc Surg. 2022 Apr;63(4):557-565. doi: 10.1016/j.ejvs.2022.02.002. Epub 2022 Feb 9. PMID 35283003